CLINICAL TRIAL: NCT03976778
Title: Evaluation of an Interventional Program for Family Physicians on Well-child Care for Children Under-5 in Suez Canal Area, Egypt
Brief Title: Evaluation of an Interventional Program for Family Physicians on Well-child Care for Children Under-5
Acronym: Well-child
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Hazem Ahmed Sayed Ahmed Sayed Ahmed, Principal investigator, Suez Canal University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Well-child care; FOM-SCU (Other: Suez Canal University)
Record Dates: First submitted 2019-05-21; First posted 2019-06-06 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Well-child Care
Keywords: Well-child; Pediatric health maintenance; Health supervision for children

STUDY DESIGN:
Intervention Model Description: A pre-post interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- a pre-post interventional study (Other): intervention consisted of 3 repeated workshops, every workshop had held for 2 days, one day per week, the number of attendants was appropriate/workshop (10 - 15).
  Interventions: Other: Training program for family physicians on well-child care for children under-5 years

INTERVENTIONS:
Other: Training program for family physicians on well-child care for children under-5 years — The researchers designed this intervention, which consisted of 3 repeated workshops, every workshop had held for 2 days, one day per week, the number of attendants was appropriate/workshop (10 - 15).

SUMMARY:
Background

Despite providing health promotion and preventive measures for children under-5 years are essential for lifelong health and wellbeing of individuals and countries, studies into family physicians' knowledge, attitudes, and practices (KAP) regarding comprehensive well-child services for children under-5 years seem to be scarce in developing countries. This study aimed to evaluate family physicians' KAP towards well-child care for children under-5 years in Suez Canal area before and after implementing an interventional program.

Methods A pre-post interventional study was conducted from September 2014 to March 2016 on comprehensive sample of 39 family physicians, who were under training in the Family Medicine department, Faculty of Medicine, Suez Canal University. Their KAP were assessed by valid and reliable questionnaire (78-items) at baseline and after 6 months of implementing a training program.

DETAILED DESCRIPTION:
A pre-post interventional study was conducted from September 2014 to March 2016. This interventional study was held in the Family Medicine Department, FOM/SCU. The assessment of participants' practices was performed in training family practice centers (FPCs) affiliated to Family Medicine Department, FOM/SCU in Port Said (2 centers), Ismailia (3 centers) and Suez governorates (4 centers).

Comprehensive sample of 39 family physicians (FPs) was recruited (the response rate was 63.93%), who accepted to participate in this intervention, affiliated to Family Medicine Department, FOM/SCU, and Ministry of Health and Population (MOHP) and regularly enrolled in classic postgraduate programs of Family Medicine Department, FOM/SCU.

The study excluded FPs who did not work in Suez Canal region despite they were under training of Family Medicine Department (FOM/SCU), were not adherent to attend the training program, did not send one of the pretest or posttest and staff of Family Medicine Department, FOM/SCU.

This study was conducted at 3 phases: preparatory, design and implementation of a training course, scoring of KAP questionnaire and evaluation and data management. During the preparatory phase; the questionnaire was designed by the researchers based on relevant literature [4,21-26].

This questionnaire consisted of 4 parts; the participants' socio-demographic data, and KAP of them towards well-child care for children under-5 years in Suez Canal area. The first 3 parts of this questionnaire were self-reported by FPs and the fourth part (practices) was assessed by the corresponding author via observational checklist during 12 months well-child visits, because of every well-child visit has its unique items of assessment in literatures and this visit included the most of targeted training practices in the present study.

Each part of questionnaire's KAP consisted of 3 subscales e.g. growth and developmental monitoring, risk assessment and screening, vaccination, chemoprevention and counseling for children under-5.

The participants' KAP were assessed by 30 multiple choice questions (MCQs), 33 items of a five-point Likert scale (with options of strongly disagree, disagree, no opinion, agree and strongly agree) and 15 items of 5-point rating scale (with options of clear unperformed, partially unperformed, borderline performed, partially performed and clear performed), respectively.

The questionnaire was validated by 3 experts in family medicine. A pilot study included 10 participants, who included in the investigator's sample size; it tested questionnaire's reliability and assessed the understandability of its items, clearness, acceptability and meaning to subjects. Cronbach's alpha was used as an internal consistency estimate of the reliability of KAP questionnaire (0.77, 0.80, and 0.81, respectively). Completion of this questionnaire lasted from 40 minutes to 50 minutes.

The percentage of correct answers of MCQs was calculated as a representative of knowledge score for each participant. While each response for Likert items was scored on a scale of 1 (strongly disagree) to 5 (strongly agree), each response for reverse-coded Likert items was re-coded and scored on a scale of 5 (strongly disagree) to 1 (strongly agree). For each individual, score of attitudes' responses was summed and converted into percentages (20-100%) to represent the attitudes score.

Each item for rating scale of practices was scored on a scale of 0 (clear unperformed) to 4 (clear performed). For each individual, score of items was summed and converted into percentage to represent the participant's practices score. The scores of knowledge and practices were considered acceptable if they were ≥ 60% according to the working bylaws in FOM/SCU. The scores of attitudes were considered positive attitudes if they were ≥ 80 %.

These data were collected at baseline and after 6 months of participation in interventional study. The researchers designed this intervention, which consisted of 3 repeated workshops, every workshop had held for 2 days, one day per week, the number of attendants was appropriate/workshop (10 - 15).

Statistical analysis Data were analyzed by SPSS version 20. Paired t test was used to compare the means of participants' KAP. The 5-point scale items of attitudes were condensed into 2 categories then McNamara's test was used to compare participants' Knowledge and attitudes changes in this study. The 5-point rating scale items of practices were condensed into 3 categories the marginal homogeneity was used to compare participants' difference of practices in this pre-post intervention.

Pearson's correlation coefficient was used to assess correlation between participants' KAP. Multiple linear regression was used to detect predictors of posttest practices score (dependent variable) and independent variables (affiliation, posttest knowledge score, duration of practice and posttest attitudes score). Stepwise linear regression was used to explore the contribution of the significant independent variables to the used model.

ELIGIBILITY:
Inclusion Criteria:

* Family physicians affiliated to MOHP and regularly enrolled in classic postgraduate programs of family medicine department, FOM, SCU within the time of the study.
* Family physicians affiliated to family medicine department (FOM, SCU) and regularly enrolled in postgraduate programs of family medicine department, FOM, SCU within the time of the study.

Exclusion Criteria:

* Family physicians exposed to similar intervention in the present and past.
* Family physicians who were under training of family medicine department (SCU), but they did not work in Suez Canal region e.g. trainee of credit hour program or FPs moved to work in other governorates within the time of the study.
* Family physicians who were not adherent to attend the training program or they did not send one of the pretest or posttest.
* Staff of family medicine department.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
to evaluate difference in total knowledge scores of participants on well-child care for under 5 years children in the pre-post intervention. | Pretest lasted 3 months and post-test questionnaire was assessed after 6 months of the interventional program
  Paired t test was used to compare the total means of participants' knowledge changes (changes in the mean percentage of the correct answers) in the pre-post intervention.
  Participants' knowledge was assessed via 30 multiple choice questions, which were designed by research team.
to evaluate changes in acceptable level of knowledge subscales in the pre-post intervention. | Pretest lasted 3 months and post-test questionnaire was assessed after 6 months of the interventional program
  Participants' Knowledge assessment included 3 subscales
  1. Growth and developmental monitoring subscale, which was assessed by nine multiple choice questions
  2. Risk assessment and screening subscale, which was assessed by eleven multiple choice questions
  3. Vaccination, chemoprevention and counseling subscale, which was assessed by ten multiple choice questions The scores of knowledge in each subscale were considered acceptable if they were ≥ 60 %, according to the regulations in Faculty of Medicine, Suez Canal University.
  McNamara's test was used to compare the knowledge's categorical changes in the pre-post intervention.
to evaluate changes in correct knowledge of participants towards well-child care in the pre-post intervention. | Pretest lasted 3 months and post-test questionnaire was assessed after 6 months of the interventional program
  Participants' Knowledge assessment included 30 multiple choice questions McNamara's test was used to compare the knowledge's categorical changes in the pre-post intervention.
to evaluate difference in total attitudes scores of participants towards well-child care for children under-5 years in Suez Canal area before and after implementing an interventional program. | Pretest lasted 3 months and post-test questionnaire was assessed after 6 months of the interventional program
  Participants' attitudes were assessed by 33-Likert items, which were arranged in a five-point Likert scale with options of "strongly disagree," "disagree," "no opinion," "agree" and "strongly agree." It included 5 attitudes-items with reverse codes.
  Each response for Likert items was scored on a scale of 1 (strongly disagree) to 5 (strongly agree).
  Each response for reverse-coded Likert items was re-coded and scored on a scale of 5 (strongly disagree) to 1 (strongly agree). For each individual, score of attitudes' responses was summed and converted into percentages (20-100 %) to represent the attitude score.
  Paired t test was used to compare the total means of participants' attitudes in the pre-post intervention.
to evaluate changes of positive attitudes subscales before and after implementing an interventional program. | Pretest lasted 3 months and post-test questionnaire was assessed after 6 months of the interventional program
  Participants' attitudes assessment included 3 subscales
  1. Growth and developmental monitoring subscale, which was assessed by 11-Likert items. Items with numbers 5 and 7 were reverse codes.
  2. Risk assessment and screening subscale, which was assessed by 9-Likert items. Items with numbers 16 and 20 were reverse codes.
  3. Vaccination, chemoprevention and counseling subscale, which was assessed by 13-Likert items. item with number 31 was reverse code.
  The scores of each attitudes subcales were considered positive attitudes if they were ≥ 80 %.
  McNamara's test was used to compare the attitudes' changes in the pre-post intervention.
to evaluate changes of positive attitudes items of participants before and after implementing an interventional program. | Pretest lasted 3 months and post-test questionnaire was assessed after 6 months of the interventional program
  The scores of attitudes were considered positive attitudes if they were ≥ 80 % (agree and strongly agree).
  The 5-point Liker scale responses were condensed into 2 categories (positive attitudes and negative attitudes) then McNamara's test was used to compare the attitudes' changes in the pre-post intervention.
to evaluate difference in total practices scores itowards well-child care for children under-5 years in Suez Canal area before and after implementing an interventional program. | Pretest lasted 3 months and post-test questionnaire was assessed after 6 months of the interventional program it also lasted 3 months.
  Family physicians' practice was assessed by the main researcher via observational checklist, which included 15 practices-items, which were arranged in a 5-point rating scale with options of "clear unperformed," "partially unperformed," "borderline performed," "partially performed" and "clear performed." The names of these options were developed by the main researcher.
  Each item for rating scale of practices was scored on a scale of 0 (clear unperformed) to 4 (clear performed). For each individual, score of items was summed and converted into percentage to represent the participant's practice score.
  Paired t test was used to compare the total means of participants' practices changes in the pre-post intervention.
to evaluate difference in acceptable level of practices subscales before and after implementing an interventional program. | Pretest lasted 3 months and post-test questionnaire was assessed after 6 months of the interventional program it also lasted 3 months.
  The scores of practices were considered acceptable if they were ≥ 60 % according to the regulations in Faculty of Medicine, Suez Canal University.
  McNamara's test was used to compare the practices' changes in each subscale in the pre-post intervention.
to evaluate changes in practices items before and after implementing an interventional program. | Pretest lasted 3 months and post-test questionnaire was assessed after 6 months of the interventional program it also lasted 3 months.
  The rating scale of practices was condensed in 3 categories clear unperformed/partially unperformed, borderline performed and partially performed/clear performed.
  Marginal homogeneity was used to compare changes in participants' practices items in the pre-post intervention.

SECONDARY OUTCOMES:
Correlation of knowledge and attitudes of participants towards well-child care for children under 5 years in the posttest | Within 4 months of ending posttest assessment.
  Pearson's correlation coefficient was used to assess correlation between total posttest score of knowledge and total posttest score of attitudes
Correlation of knowledge and practices of participants towards well-child care for children under 5 years in the posttest | Within 4 months of ending posttest assessment.
  Pearson's correlation coefficient was used to assess correlation between total posttest score of knowledge and total posttest score of practices
Correlation of attitudes and practices of participants towards well-child care for children under 5 years in the posttest | Within 4 months of ending posttest assessment.
  Pearson's correlation coefficient was used to assess correlation between total posttest score of attitudes and total posttest score of practices
Predictors of posttest practices of participants towards well-child care for children under 5 years. | Within 4 months of ending posttest assessment.
  Multiple linear regression was used to detect predictors of posttest practice score (dependent or outcome variable) and independent variables (affiliation, posttest knowledge score and duration of practice).

CONTACTS AND LOCATIONS:
Overall Officials: Hazem A Sayed Ahmed, PhD, Principal Investigator — Family medicine Department, Faculty of Medicine, Suez Canal University, Egypt
Locations (1):
- Faculty of Medicine, Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
SPSS documents
Supporting Information: ICF
Time Frame: After acceptance of publication and getting permission from the main author The data will be available for years
Access Criteria: Links of journal which accept the manuscript for publication